CLINICAL TRIAL: NCT01974349
Title: A Phase I, Randomized, Open-label, Single-center, Crossover Study to Assess the Effect of Food on the Pharmacokinetics of a 75 mg Single Oral Dose of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Male Volunteers Aged 18 to 45 Years
Brief Title: To Assess the Effect of Food on the Pharmacokinetics of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00069
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Solid Tumours
Keywords: Phase I, healthy, pharmacokinetics, food effect.
MeSH Terms: interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- selumetinib 75mg (oral capsule fasted) (Experimental): Volunteers will recieve selumetinib 75mg administered by mouth, as a capsule, in a fasted state.
  Interventions: Drug: selumetinib (oral)
- selumetinib 75mg (oral capusle fed) (Experimental): Volunteers will receive selumetinib 75mg administered by mouth, as a capsule, in a fed state.
  Interventions: Drug: selumetinib (oral)

INTERVENTIONS:
Drug: selumetinib (oral) — Volunteers will receive: 75 mg selumetinib oral dose in a fasted state (Treatment A) followed by a second 75 mg selumetinib oral dose in the fed state (Treatment B) with a washout period of at least 7 days between doses, or: 75 mg selumetinib oral dose in the fed state (Treatment B) followed by a second 75 mg selumetinib oral dose in the fasted state (Treatment A) with a washout period of at least 7 days between doses.
  Other Names: AZD6244

SUMMARY:
Study to assess the effect of food on the Pharmacokinetics of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Male Volunteers

DETAILED DESCRIPTION:
A randomized, Open-label, Single-center, Crossover Study to Assess the Effect of Food on the Pharmacokinetics of a 75 mg Single Oral Dose of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria: 1. Have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive). 2. Must not have smoked or used nicotine products within the previous 3 months. 3. Have a calculated creatinine clearance (CrCL) greater than 50 mL/min using the Cockcroft-Gault formula.

Exclusion Criteria: 1. Current or past history of central serous retinopathy or retinal vein thrombosis, intra-ocular pressure greater than 21 mmHg or uncontrolled glaucoma. 2. Any clinically relevant abnormal findings in physical examination, hematology, clinical chemistry, urinalysis, vital signs, or ECG at baseline in the opinion of the investigator. 3. History or presence of any clinically significant disease or disorder in the opinion of the investigator. 4. Subjects of Japanese or non-Japanese Asian ethnicity. 5. Subjects where any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese Asian (e.g., China, Taiwan, Korea, Philippines, Thailand, Vietnam and Malaysia). Asian Indians are acceptable.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of selumetinib and N desmethyl selumetinib, by assessment of maximum plasma concentration (Cmax) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments

SECONDARY OUTCOMES:
Pharmacokinetics of selumetinib and N desmethyl selumetinib, by assessment of the area under the plasma concentration-time curve from time zero to infinity (AUC) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib, by assessment of the area under the plasma concentration-time curve from time zero to the time of the last measurable concentration AUC(0-t) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib, by assessment of area under the plasma concentration-time curve from time zero to 12 hours postdose AUC (0-12) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib, by assessment of time to Cmax (tmax) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib by assessment of apparent systemic plasma clearance (CL/F) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib by assessment of apparent volume at distribution equilibrium, mean residence time (MRT)*CL/F (Vss/F) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib by assessment of apparent volume at distribution (Vz/F) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib by assessment of terminal half-life (t½) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib by assessment of terminal rate constant (λz) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib by assessment of (MRT) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib by assessment of AUC metabolite to parent ratio, N-desmethyl selumetinib AUC/selumetinib (AUC MRAUC) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments
Pharmacokinetics of selumetinib and N desmethyl selumetinib by assessment of Cmax metabolite to parent ratio, N-desmethyl selumetinib Cmax/selumetinib Cmax (MRCmax) | Blood samples are collected pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, and 48 hours postdose
  Curve taken during each of the 2 treatments

OTHER OUTCOMES:
Safety variables (adverse events, physical examinations, ophthalmologic assessments, vital signs, clinical laboratory assessments, and 12 lead electrocardiograms) | Baseline (Day-1) up to Day 24
  Assessments performed during each of the 2 treatments

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, Principal Investigator — Quintiles 6700 W 115th Street, Kansas, US
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Tomkinson H, McBride E, Martin P, Lisbon E, Dymond AW, Cantarini M, So K, Holt D. Comparison of the Pharmacokinetics of the Phase II and Phase III Capsule Formulations of Selumetinib and the Effects of Food on Exposure: Results From Two Randomized Crossover Trials in Healthy Male Subjects. Clin Ther. 2017 Nov;39(11):2260-2275.e1. doi: 10.1016/j.clinthera.2017.08.022. Epub 2017 Oct 4. PMID 28985960